CLINICAL TRIAL: NCT01797718
Title: Constitutional Delay of Growth and Puberty: Towards Evidence-based Treatment
Acronym: CDGP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Foundation for Paediatric Research, Finland (Other)
Responsible Party: Principal Investigator, Tero Varimo, MD, PhD, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT:2012-002477-59
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Constitutional Delay of Growth and Puberty
Keywords: Puberty; Constitutional; Delay; Letrozole; Testosterone
MeSH Terms: interventions — Testosterone; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone (Active Comparator): ~1mg/kg every 4 weeks for 6 months
  Interventions: Drug: Testosterone
- Letrozole (Active Comparator): 2.5mg daily for 6 months
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Testosterone — 1mg/kg every 4 weeks for 6 months
  Other Names: Sustanon 250
  Arms: Testosterone
Drug: Letrozole — 2.5mg daily for 6 months. Safety criteria: if testosterone level is above 30nM at 3 months, the dosage is reduced to 2.5mg every other day
  Other Names: Letrozole Bluefish; Letrozole Orion; Letrozole Accord; Letrozole Sandoz; Femar
  Arms: Letrozole

SUMMARY:
Boys with constitutional delay of growth and puberty (CDGP) should be offered evidence-based effective and safe treatment option. This study compares the effects of low-dose testosterone and aromatase inhibitor letrozole on pubertal progression. The hypothesis is that, in boys CDGP showing earliest signs of puberty, peroral letrozole (2.5 mg/d for 6 mo) induces faster biochemical and clinical progression of puberty as compared to low-dose intramuscular testosterone Rx (~1mg/kg/mo for 6 mo). In addition, 10 or more boys who select watchful waiting instead of medication will provide background data on the natural progression of CDGP, and their data will not be used in primary statistical comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Constitutional delay of growth and puberty
* Age 14 years or more
* mean testicular volume 2.5 ml or more and less than 4 ml
* serum testosterone level less than 5 nM OR

as above, but serum testosterone 1 nM or more with normal DHEAS level, even if the mean testicular volume is less than 2.5 ml OR

as above, but tanner stage G2 and testosterone level less than 3 nM

Exclusion Criteria:

* Chronic diseases
* Primary or secondary hypogonadism
* Chromosomal anomalies
* Chronic medication that potentially adversely affects bone mineralization (excluding inhaled corticosteroid treatment)

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
testicular volume | one year
  Testes will be measured with a ruler to the nearest millimeter and volume will be calculated at 0, 6, and 12 mo
clinical and biochemical measures of pubertal progression | one year
  Activity of the hypothalamic-pituitary-gonadal axis, evaluated by
  * genital and pubic hair stage of puberty according to Tanner;
  * growth velocity (cm/yr);
  * basal and gonadotropin-releasing hormone (GnRH)-stimulated gonadotropin levels;
  * urinary luteinizing hormone levels;
  * testosterone;
  * inhibin B;
  * anti-mullerian hormone (AMH)

SECONDARY OUTCOMES:
Bone health | one year
  Several endpoints related to bone health
Psychosocial well-being | one year
  Psycho-social well-being will assessed with questionnaires.
Puberty-related metabolical and clinical changes | one year
  Biochemical and metabolical changes will be compared btw testosterone and letrozole treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Taneli Raivio, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Matti Hero, MD, PhD, Study Director — Helsinki University Central Hospital; Tero Varimo, MD, PhD, Study Chair — Helsinki University Central Hospital; Päivi Miettinen, MD, PhD, Study Chair — Helsinki University Central Hospital; Jorma Toppari, MD, PhD, Study Chair — University of Turku; Hanna Huopio, MD, PhD, Study Chair — Kuopio University Central Hospital; Sirpa Tenhola, MD, PhD, Study Chair — Kymeenlaakso Central Hospital; Raimo Voutilainen, MD, PhD, Study Chair — Kuopio University Central Hospital
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Kotka Central Hospital, Kotka
  - Kuopio University Central Hospital, Kuopio
  - Turku University Central Hospital, Turku

REFERENCES:
- [Derived] Varimo T, Miettinen PJ, Huopio H, Rikkonen T, Voutilainen R, Tenhola S, Raivio T, Hero M. Impact of aromatase inhibition on bone mineral density and structure: a randomized controlled trial in boys with delayed puberty. Eur J Endocrinol. 2025 Jul 31;193(2):289-296. doi: 10.1093/ejendo/lvaf160. PMID 40796279
- [Derived] Kariola L, Varimo T, Huopio H, Tenhola S, Voutilainen R, Kosola S, Toppari J, Sintonen H, Miettinen PJ, Raivio T, Hero M. Health-related quality of life in boys with constitutional delay of growth and puberty. Front Endocrinol (Lausanne). 2022 Nov 25;13:1028828. doi: 10.3389/fendo.2022.1028828. eCollection 2022. PMID 36518253
- [Derived] Huttunen H, Varimo T, Huopio H, Voutilainen R, Tenhola S, Miettinen PJ, Raivio T, Hero M. Serum testosterone and oestradiol predict the growth response during puberty promoting treatment. Clin Endocrinol (Oxf). 2022 Feb;96(2):220-226. doi: 10.1111/cen.14605. Epub 2021 Oct 1. PMID 34596269
- [Derived] Kohva E, Varimo T, Huopio H, Tenhola S, Voutilainen R, Toppari J, Miettinen PJ, Vaaralahti K, Viinamaki J, Backman JT, Hero M, Raivio T. Anti-Mullerian hormone and letrozole levels in boys with constitutional delay of growth and puberty treated with letrozole or testosterone. Hum Reprod. 2020 Feb 29;35(2):257-264. doi: 10.1093/humrep/dez231. PMID 31958337
- [Derived] Varimo T, Huopio H, Kariola L, Tenhola S, Voutilainen R, Toppari J, Toiviainen-Salo S, Hamalainen E, Pulkkinen MA, Laaperi M, Tarkkanen A, Vaaralahti K, Miettinen PJ, Hero M, Raivio T. Letrozole versus testosterone for promotion of endogenous puberty in boys with constitutional delay of growth and puberty: a randomised controlled phase 3 trial. Lancet Child Adolesc Health. 2019 Feb;3(2):109-120. doi: 10.1016/S2352-4642(18)30377-8. Epub 2019 Jan 4. PMID 30612946